CLINICAL TRIAL: NCT03169452
Title: Clinical Application and Outcome of Non-invasive Ventilation in Different Chest Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, principal investigator, Assiut University
Other Study IDs: NIV
Record Dates: First submitted 2017-05-25; First posted 2017-05-30 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Chest--Diseases
MeSH Terms: interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Non-invasive mechanical ventilator — mechanical assisted breaths without the placement of an artificial way
  Other Names: continuous positive airway pressure

SUMMARY:
Noninvasive ventilation is increasingly used method of respiratory management in both the emergency room and critical care. Noninvasive ventilation delivers mechanically assisted breaths without the placement of an artificial airway and has become an important mechanism of ventilator support inside and outside the intensive care unit.

Noninvasive ventilation is further subdivided into negative pressure ventilation which is the iron lung, first used in 1928 and the Hayek oscillator, is a more recently designed to provide negative pressure during inspiration and positive pressure during expiration. Noninvasive positive pressure ventilation can be used as continuous positive airway pressure or bi-level positive airway pressure.

ELIGIBILITY:
Inclusion Criteria:

* obstructive sleep apnea syndrome
* acute exacerbation Chronic obstructive pulmonary disease
* pneumonia
* interstitial lung diseases

Exclusion Criteria:

* Patients refuse Non invasive ventilation
* Patients with absolute indication for Mechanical ventilator (in respiratory arrest or unstable cardiorespiratory status, trauma or burns involving the face, or gastric surgery, reduced consciousness, Pneumothorax
* Patients with contraindication to Non invasive ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who admitted to the Respiratory intensive care unit and the attending team conducted him to Non invasive ventilation
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
percentage of patients need mechanical ventilation | 1-48 hours
  the number of patients without improvement on non-invasive ventilator and require transfer to mechanical ventilator

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No